CLINICAL TRIAL: NCT00289783
Title: A Phase III, Randomized, Multinational Study, Double-blinded for the Immunogenicity and Consistency Evaluation of 3 Hib-MenCY-TT Vaccine Lots and Single-blinded and Controlled for the Evaluation of Safety and Immunogenicity of GSK Biologicals' Haemophilus Influenzae Type b and Neisseria Meningitidis Serogroups C and Y-tetanus Toxoid Conjugate Vaccine Combined (Hib-MenCY-TT) Compared to Monovalent Hib Vaccine in Healthy Infants at 2, 4, 6, and 12 to 15 Months of Age.
Brief Title: Safety and Immunogenicity Study of Hib-MenCY-TT Vaccine Compared to Licensed Hib Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 103813; 105067 (Other: GSK)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2012-08-06 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2016-11

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
Keywords: Primary and booster vaccination; Neisseria meningitidis; Hib disease; Meningococcal vaccine; Meningococcal disease; Children; Immunogenicity; Safety; Infants
MeSH Terms: conditions — Haemophilus Infections; Meningococcal Infections | interventions — Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; Haemophilus influenzae-type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine; PEDIARIX; Heptavalent Pneumococcal Conjugate Vaccine; Measles-Mumps-Rubella Vaccine; Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- Menhibrix A Group (Experimental): Subjects were primed with 3 doses of Menhibrix vaccine Lot A co-administered with Pediarix and boosted with 1 dose of Menhibrix vaccine, with co-administration of M-M-R II and Varivax. Subjects received vaccination at approximately 2, 4, 6 months and the fourth dose at 12-15 months of age. Menhibrix and Pediarix vaccines were administered intramuscularly in the right or left upper thigh, respectively. M-M-R II and Varivax vaccines were administered subcutaneously respectively in the upper left arm and the upper right arm.
  Interventions: Biological: GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis 792014 vaccine; Biological: Pediarix; Biological: Prevnar; Biological: M-M-R II; Biological: Varivax
- Menhibrix B Group (Experimental): Subjects were primed with 3 doses of Menhibrix vaccine Lot B co-administered with Pediarix and boosted with 1 dose of Menhibrix vaccine, with co-administration of M-M-R II and Varivax. Subjects received vaccination at approximately 2, 4, 6 months and the fourth dose at 12-15 months of age. Menhibrix and Pediarix vaccines were administered intramuscularly in the right or left upper thigh, respectively. M-M-R II and Varivax vaccines were administered subcutaneously respectively in the upper left arm and the upper right arm.
  Interventions: Biological: GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis 792014 vaccine; Biological: Pediarix; Biological: Prevnar; Biological: M-M-R II; Biological: Varivax
- Menhibrix C Group (Experimental): Subjects were primed with 3 doses of Menhibrix vaccine Lot C co-administered with Pediarix and boosted with 1 dose of Menhibrix vaccine, with co-administration of M-M-R II and Varivax. Subjects received vaccination at approximately 2, 4, 6 months and the fourth dose at 12-15 months of age. Menhibrix and Pediarix vaccines were administered intramuscularly in the right or left upper thigh, respectively. M-M-R II and Varivax vaccines were administered subcutaneously respectively in the upper left arm and the upper right arm.
  Interventions: Biological: GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis 792014 vaccine; Biological: Pediarix; Biological: Prevnar; Biological: M-M-R II; Biological: Varivax
- Menhibrix Group (Experimental): Subjects were primed with 3 doses of Menhibrix vaccine Lot A, B or C co-administered with Pediarix and boosted with 1 dose of Menhibrix vaccine, with co-administration of M-M-R II and Varivax. Subjects received vaccination at approximately 2, 4, 6 months and the fourth dose at 12-15 months of age. Menhibrix and Pediarix vaccines were administered intramuscularly in the right or left upper thigh, respectively. M-M-R II and Varivax vaccines were administered subcutaneously respectively in the upper left arm and the upper right arm.
  Interventions: Biological: GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis 792014 vaccine; Biological: Pediarix; Biological: Prevnar; Biological: M-M-R II; Biological: Varivax
- ActHIB Group (Active Comparator): Subjects were primed with 3 doses of ActHIB co-administered with Pediarix and boosted with 1 dose of PedvaxHIB, with co-administration of M-M-R II and Varivax. Subjects received vaccination at approximately 2, 4, 6 months and the fourth dose at 12-15 months of age. ActHIB, PedvaxHIB vaccines were administered intramuscularly in the right upper thigh and Pediarix vaccine in the left upper thigh. M-M-R II and Varivax vaccines were administered subcutaneously respectively in the upper left arm and the upper right arm.
  Interventions: Biological: ActHIB; Biological: PedvaxHIB

INTERVENTIONS:
Biological: GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis 792014 vaccine — 3-dose intramuscular injection at 2, 4 and 6 months of age, and 1 booster dose by intramuscular injection at 12 to 15 months of age.
  Arms: Menhibrix A Group; Menhibrix B Group; Menhibrix C Group; Menhibrix Group
Biological: ActHIB — 3-dose intramuscular injection at 2, 4 and 6 months of age.
  Arms: ActHIB Group
Biological: PedvaxHIB — 1 booster dose by intramuscular injection at 12 to 15 months of age.
  Arms: ActHIB Group
Biological: Pediarix — 3-dose intramuscular injection at 2, 4 and 6 months of age.
  Other Names: Infanrix penta
  Arms: Menhibrix A Group; Menhibrix B Group; Menhibrix C Group; Menhibrix Group
Biological: Prevnar — 3-dose intramuscular injection at 2, 4 and 6 months of age, and 1 booster dose by intramuscular injection at 12 to 15 months of age.
  Arms: Menhibrix A Group; Menhibrix B Group; Menhibrix C Group; Menhibrix Group
Biological: M-M-R II — 1 booster dose by subcutaneous injection at 12 to 15 months of age.
  Arms: Menhibrix A Group; Menhibrix B Group; Menhibrix C Group; Menhibrix Group
Biological: Varivax — 1 booster dose by subcutaneous injection at 12 to 15 months of age
  Arms: Menhibrix A Group; Menhibrix B Group; Menhibrix C Group; Menhibrix Group

SUMMARY:
This study evaluates the immunogenicity and consistency of 3 Hib-MenCY-TT vaccine lots and the safety and immunogenicity of Hib-MenCY-TT vaccine compared to a control group receiving licensed Hib conjugate vaccine, when each are co-administered with Pediarix® to healthy infants at 2, 4, and 6 months of age. The study will also evaluate the safety and immunogenicity of Hib-MenCY-TT vaccine compared to a control group receiving licensed Hib conjugate vaccine, when each are co-administered with M-M-R® II and Varivax® at 12 to 15 months of age.

DETAILED DESCRIPTION:
The subjects from this study will participate in one of three cohorts:

* US Safety and Immunogenicity (Cohort 1): All immunogenicity analyses in the primary and booster phases will be evaluated in this cohort. These subjects will also contribute to the safety analyses in the primary and booster phases.
* Safety Only (Cohort 2): Only safety objectives will be assessed in the primary and booster phases for this cohort.
* Non-US Safety and Immunogenicity (Cohort 3): Only descriptive immunogenicity results in the primary and booster phases will be reported for this cohort. These subjects will also contribute to the safety analyses in the primary and booster phases.

Treatment allocation:

Primary phase: Subjects will be randomized with balanced allocation (1:1:1:1) to 1 of the 4 treatment groups and with a stratification according to the cohort. Assignment to a cohort will be based on study site.

Booster phase: Subjects who received Hib-MenCY-TT vaccine in the primary phase will receive a booster dose of Hib-MenCY-TT vaccine. Subjects who received ActHIB in the primary phase will receive a booster dose of PedvaxHIB.

During the 3-dose primary vaccination course, co-administration of Prevnar, Synagis, and/or rotavirus vaccine is permitted; co-administration of influenza vaccine is permitted at dose 3.

During the booster vaccination, co-administration of Prevnar, hepatitis A vaccine and influenza vaccine is permitted for all subjects in Cohort 1, 2 and 3; and co-administration of measles, mumps, rubella and varicella vaccine is permitted for all subjects in Cohort 2 and 3.

The study will be conducted in a double-blind fashion with regard to consistency of the 3 manufacturing lots of Hib-MenCY-TT vaccine and single-blind fashion for Hib-MenCY-TT vaccine versus monovalent Hib vaccine. The parents/guardians will be blinded up to collection of all data pertaining to the period up to one month after booster vaccination. Therefore, the extended safety follow-up after the booster dose will be conducted in an unblinded manner. The person administering the vaccines will ensure that the parent/guardian does not see the vaccine vial used in reconstituting the vaccine. Due to the differences in the presentations of the candidate Hib-MenCY-TT vaccine and control vaccines, it is not possible to blind study personnel who administer the vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes that parents/guardians can and will comply with the requirements of the protocol
* A male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after 36 weeks gestation.
* Infants who have not received a previous dose of hepatitis B vaccine or those who have received only 1 dose of hepatitis B vaccine administered at least 30 days prior to enrollment.
* Infants may have received a birth dose of Bacillus Calmette-Guérin (BCG) vaccine.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of study vaccine(s). (Synagis® [palivizumab, MedImmune], Prevnar (Prevenar), rotavirus vaccine, and influenza vaccine are allowed.
* Previous vaccination against Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, and/or poliovirus; more than one previous dose of hepatitis B vaccine.
* History of Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, hepatitis B, and/or poliovirus disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing is required).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including dry natural latex rubber.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at time of enrollment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Concurrent participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).

Additional specific criteria for the US subjects in Cohort 1. In addition, for Cohorts 2 and 3, subjects should not be administered M-M-R II and Varivax if any of these criteria apply:

* History of measles, mumps, rubella or varicella.
* Previous vaccination against measles, mumps, rubella or varicella.
* Hypersensitivity to any component of the vaccines, including gelatin or neomycin.
* Patients receiving immunosuppressive therapy.
* Individuals with blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* Individuals with primary and acquired immunodeficiency states.
* Individuals with a family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* Individuals with active tuberculosis.
* Acute disease at time of booster vaccination.

Ages: 6 Weeks to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4441 (Actual)
Dates: Start 2006-02-22; Primary Completion 2007-08-27 (Actual); Study Completion 2008-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (84):
- United States (79):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bryant, Arkansas
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, East Artesia, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Cocoa Beach, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Rockledge, Florida
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Jamaica Plain, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Brainerd, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, North Las Vegas, Nevada
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, New Hartford, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Sylva, North Carolina
  - GSK Investigational Site, Boardman, Ohio
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Huber Heights, Ohio
  - GSK Investigational Site, South Euclid, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Beaver Falls, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Lexington, South Carolina
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Pleasant Grove, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, Mechanicsville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, La Crosse, Wisconsin
- Australia (4):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Carlton, Victoria
- GSK Investigational Site, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bryant KA, Marshall GS. Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine for infants and toddlers. Expert Rev Vaccines. 2011 Jul;10(7):941-50. doi: 10.1586/erv.11.90. PMID 21806393
- [Background] Bryant KA, Marshall GS, Marchant CD, Pavia-Ruiz N, Nolan T, Rinderknecht S, Blatter M, Aris E, Lestrate P, Boutriau D, Friedland LR, Miller JM. Immunogenicity and safety of H influenzae type b-N meningitidis C/Y conjugate vaccine in infants. Pediatrics. 2011 Jun;127(6):e1375-85. doi: 10.1542/peds.2009-2992. Epub 2011 May 29. PMID 21624883
- [Background] Bryant K, McVernon J, Marchant C, Nolan T, Marshall G, Richmond P, Marshall H, Nissen M, Lambert S, Aris E, Mesaros N, Miller J. Immunogenicity and safety of measles-mumps-rubella and varicella vaccines coadministered with a fourth dose of Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine in toddlers: a pooled analysis of randomized trials. Hum Vaccin Immunother. 2012 Aug;8(8):1036-41. doi: 10.4161/hv.20357. Epub 2012 Aug 1. PMID 22617844
- [Background] Bryant KA et al. Immune response to measles, mumps, rubella (MMR) and varicella (V) vaccine coadministered with a fourth dose of Haemophilus influenzae type b - Neisseria meningitidis serogroups C and Y - tetanus toxoid conjugate (HibMenCY) vaccine in toddlers. Abstract presented at the Annual meeting of Pediatric Academic Societies (PAS). Vancouver, Canada, 1-4 May 2010.
- [Derived] Rinderknecht S, Bryant K, Nolan T, Pavia-Ruz N, Doniz CA, Weber MA, Cohen C, Aris E, Mesaros N, Miller JM. The safety profile of Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine (HibMenCY). Hum Vaccin Immunother. 2012 Mar;8(3):304-11. doi: 10.4161/hv.18752. Epub 2012 Feb 13. PMID 22327493
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 103813 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103813 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103813 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103813 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103813 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 103813 are summarised with study 105067 on the GSK Clinical Study Register.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized at the beginning of the primary phase and kept their group assignment during the fourth dose vaccination phase. The study protocol identified 3 different study cohorts : United States (US) Safety and Immunogenicity (Cohort 1), Safety Only (Cohort 2: from all investigation sites), Non-US Safety and Immunogenicity (Cohort 3).
Pre-assignment Details: The data for 261 subjects from one study center in the US were not included in the analyses as vaccine accountability could not be fully reconciled (i.e. treatment group assignment for the different subjects could not be verified).
Period: Primary Phase
Arm/Group | Menhibrix Group | ActHIB Group
Started | 3136 | 1044
Completed | 2888 | 961
Not Completed | 248 | 83
Not completed — Adverse Event | 10 | 1
Not completed — Protocol Violation | 27 | 6
Not completed — Withdrawal by Subject | 93 | 40
Not completed — Lost to Follow-up | 60 | 14
Not completed — Migration from the study area | 26 | 10
Not completed — Other | 32 | 12
Period: Fourth Dose Phase
Arm/Group | Menhibrix Group | ActHIB Group
Started | 2769 | 923
Completed | 2682 | 899
Not Completed | 87 | 24
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 10 | 1
Not completed — Lost to Follow-up | 53 | 12
Not completed — Migration from the study area | 1 | 1
Not completed — Other | 22 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menhibrix Group | ActHIB Group | Total
Number analyzed (Participants) | 3136 | 1044 | 4180
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.11 (0.26) | 2.11 (0.27) | 2.11 (0.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1523 | 498 | 2021
  Male | 1613 | 546 | 2159

OUTCOME MEASURES:

1. Primary Outcome: Anti-Polyribosyl Ribitol Phosphate (PRP) Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in microgram per millilitre (µg/mL)
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after primary vaccination
Population: The Primary According-To-Protocol (ATP) cohort for immunogenicity included all evaluable subjects (i.e. those who met eligibility criteria, complied with the procedures defined in the protocol and met no elimination criteria during the study) for whom results were available for antibodies against the vaccine antigens after the third vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (µg/mL)
Arm/Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 162 | 180 | 176 | 518 | 171
microgram per milliliter (µg/mL) | 10.170 [8.855 to 11.681] | 11.424 [9.710 to 13.441] | 11.438 [9.503 to 13.768] | 11.021 [10.027 to 12.114] | 6.463 [5.288 to 7.900]
Statistical Analysis 1: Comparison: Menhibrix A Group vs Menhibrix B Group; To demonstrate the lot-to-lot consistency of 3 manufacturing lots of Hib-MenCY-TT vaccine co-administered with DTPa-HBV-IPV vaccine following 3 primary doses in terms of immunogenicity for polyribosylribitol phosphate (PRP) as measured by ELISA; Test type: Equivalence — Criteria for lot-to-lot consistency (1 month after primary vaccination): For each pair of lots and for the immune response to anti-PRP measured by Enzyme Linked Immunosorbent Assay (ELISA) the two-sided 95% confidence interval (CI) on the geometric mean concentrations (GMCs) ratio between lots is within the [0.5; 2.0] interval; GMC ratio = 1.12, 95% CI 2-sided [0.89 to 1.42]
Statistical Analysis 2: Comparison: Menhibrix A Group vs Menhibrix C Group; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Criteria for lot-to-lot consistency (1 month after primary vaccination): For each pair of lots and for the immune response to anti-PRP measured by ELISA the two-sided 95% confidence interval (CI) on the geometric mean concentrations (GMCs) ratio between lots is within the [0.5; 2.0] interval; GMC ratio = 1.12, 95% CI 2-sided [0.89 to 1.42]
Statistical Analysis 3: Comparison: Menhibrix B Group vs Menhibrix C Group; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMC ratio = 1, 95% CI 2-sided [0.8 to 1.26]

2. Primary Outcome: Neisseria Meningitidis Serogroup C (MenC) Serum Bactericidal Assay Using Human Complement (hSBA) Antibody Titers
Description: Titers were expressed as Geometric Mean Titers (GMTs)
  This analysis occured on the cohort 1 : Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 158 | 168 | 165 | 491 | 164
Titers | 910.0 [754.6 to 1097.3] | 1118.0 [931.1 to 1342.5] | 885.7 [712.4 to 1101.2] | 967.6 [864.0 to 1083.5] | 2.5 [2.2 to 2.9]
Statistical Analysis 1: Comparison: Menhibrix A Group vs Menhibrix B Group; To demonstrate the lot-to-lot consistency of 3 manufacturing lots of Hib-MenCY-TT vaccine co-administered with DTPa-HBV-IPV vaccine following 3 primary doses in terms of immunogenicity for N. meningitidis serogroup C (MenC) as measured by a serum bactericidal assay using human complement (hSBA); Test type: Equivalence — For each pair of lots and for the immune response to hSBA-MenC, the two-sided 95% confidence interval (CI) on the geometric mean titers (GMTs) ratio between lots is within the [0.5; 2.0] interval; GMT ratio = 1.23, 95% CI 2-sided [0.93 to 1.62]
Statistical Analysis 2: Comparison: Menhibrix A Group vs Menhibrix C Group; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; GMT ratio = 0.97, 95% CI 2-sided [0.74 to 1.29]
Statistical Analysis 3: Comparison: Menhibrix B Group vs Menhibrix C Group; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; GMT ratio = 0.79, 95% CI 2-sided [0.6 to 1.04]

3. Primary Outcome: Neisseria Meningitidis Serogroup Y (MenY) Serum Bactericidal Assay Using Human Complement (hSBA) Antibody Titers
Description: Titers are expressen as Geometric Mean Titers (GMTs)
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 150 | 168 | 163 | 481 | 162
Titers | 178.9 [136.4 to 234.6] | 288.1 [232.8 to 356.6] | 249.6 [195.6 to 318.7] | 236.6 [205.7 to 272.1] | 2.2 [2.0 to 2.4]
Statistical Analysis 1: Comparison: Menhibrix A Group vs Menhibrix B Group; To demonstrate the lot-to-lot consistency of 3 manufacturing lots of Hib-MenCY-TT vaccine co-administered with DTPa-HBV-IPV vaccine following 3 primary doses in terms of immunogenicity for N. meningitidis serogroup Y (MenY) as measured by a serum bactericidal assay using human complement (hSBA); Test type: Equivalence — For each pair of lots and for the immune response to hSBA-MenY, the two-sided 95% confidence interval (CI) on the geometric mean titers (GMTs) ratio between lots is within the [0.5; 2.0] interval; GMT ratio = 1.61, 95% CI 2-sided [1.14 to 2.27]
Statistical Analysis 2: Comparison: Menhibrix A Group vs Menhibrix C Group; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.4, 95% CI 2-sided [0.99 to 1.97]
Statistical Analysis 3: Comparison: Menhibrix B Group vs Menhibrix C Group; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 0.87, 95% CI 2-sided [0.62 to 1.21]

4. Primary Outcome: hSBA-MenC Antibody Titers
Description: Titers are expressed as Geometric Mean Titers (GMTs)
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: Prior to the fourth dose vaccination and 42 days after the fourth dose
Population: The Fourth dose ATP cohort for immunogenicity included all evaluable subjects (i.e. those who met eligibility criteria, complied with the procedures defined in the protocol, with no elimination criteria during the study) for whom results were available for antibodies against vaccine antigens for the blood sample taken 43 days post-vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 331 | 119
Titers
  hSBA-MenC [post-dose 4] | 2039.8 [1746.3 to 2382.6] | 4.3 [3.2 to 5.8]
  hSBA-MenC [pre-dose 4]: number analyzed (Participants) | 329 | 104
  hSBA-MenC [pre-dose 4] | 180.3 [155.6 to 208.8] | 3.0 [2.4 to 3.7]
Statistical Analysis 1: Comparison: Menhibrix Group; To evaluate the specific effect of a fourth dose of Menhibrix vaccine co-administered with M-M-R II and Varivax vaccines at 12 to 15 months of age in terms of a fourth dose vaccine response as measured by hSBA-MenC; Test type: Non-Inferiority — Criteria for immunogenicity of MenC (42 days after the fourth dose): Lower limit of the asymptotic 95% CI for the geometric mean of individual ratio of post-dose 4/pre-dose 4 is ≥ 2; GMT ratio = 12, 95% CI 2-sided [10.4 to 13.8]
Statistical Analysis 2: Comparison: ActHIB Group; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Point estimate = Lower limit (LL) = Upper limit (UL) as LL and UL values were not available due to the departure from lognormal distribution (large number of imputed values); GMT ratio = 1.4, 95% CI 2-sided [1.4 to 1.4]

5. Primary Outcome: hSBA-MenY Antibody Titers
Description: as for outcome 4
Time Frame: Prior to the fourth dose vaccination and 42 days after the fourth dose
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 342 | 120
Titers
  hSBA-MenY [post-dose 4] | 1389.5 [1205.0 to 1602.2] | 48.6 [31.9 to 74.0]
  hSBA-MenY [pre-dose 4]: number analyzed (Participants) | 329 | 103
  hSBA-MenY [pre-dose 4] | 119.1 [101.1 to 140.3] | 2.5 [2.1 to 2.9]
Statistical Analysis 1: Comparison: Menhibrix Group; To evaluate the specific effect of a fourth dose of Menhibrix vaccine co-administered with M-M-R II and Varivax vaccines at 12 to 15 months of age in terms of a fourth dose vaccine response as measured by hSBA-MenY; Test type: Non-Inferiority — Criteria for immunogenicity of MenY (42 days after the fourth dose): Lower limit of the asymptotic 95% CI for the geometric mean of individual ratio of post-dose 4/pre-dose 4 is ≥ 2; GMT ratio = 11.8, 95% CI 2-sided [10.2 to 13.8]
Statistical Analysis 2: Comparison: ActHIB Group; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; GMT ratio = 21.1, 95% CI 2-sided [21.1 to 21.1]

6. Primary Outcome: Number of Subjects With Anti-PRP Antibody Concentration Equal to or Above 1.0 Microgram Per Milliliter (µg/mL)
Description: This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 162 | 180 | 176 | 518 | 171
Participants | 158 | 175 | 166 | 499 | 156

7. Primary Outcome: Number of Subjects With hSBA-MenC Titer Equal to or Above 1:8
Description: as for outcome 6
Time Frame: 42 days after the fourth dose
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 331 | 119
Participants | 326 | 26

8. Primary Outcome: Number of Subjects With hSBA-MenY Titer Equal to or Above 1:8
Description: as for outcome 6
Time Frame: 42 days after the fourth dose
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 342 | 120
Participants | 338 | 87

9. Primary Outcome: Number of Subjects With Anti-measles Antibody Concentrations Equal to or Above 150 Milli-international Units Per Milli-liter (mIU/ML)
Description: The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-measles antibody concentrations below 150 mIU/mL.
  Co-administration with MMR-II vaccine
Time Frame: 42 days after the fourth dose
Population: The Pooled cohort consisted of all evaluable subjects in the Fourth dose ATP cohort for immunogenicity, HibMenCY-TT-008 and Cohort 1 from HibMenCY-TT-010.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 852 | 286
Participants | 815 | 274
Statistical Analysis 1: Comparison: Menhibrix Group vs ActHIB Group; To demonstrate the non-inferiority of M-M-R II vaccine when co-administered with a fourth dose of Menhibrix vaccine compared to M-M-R II vaccine co-administered with a fourth dose of PedvaxHIB vaccine, each co-administered with Varivax vaccine; Test type: Non-Inferiority — Lower limit of the standardized asymptotic 95% CI for the difference (Menhibrix vaccine fourth dose group minus ActHIB fourth dose group) in the percentage of subjects with seroconversion ≥ 150 mIU/mL, in initially seronegative subjects (<150 mIU/mL), for anti-measles antibody is ≥-5% (clinical limit for non-inferiority); Difference in percentage = -0.15, 95% CI 2-sided [-2.56 to 3.06]

10. Primary Outcome: Number of Subjects With Anti-PRP Antibody Concentration Equal to or Above 1.0 Microgram Per Milliliter
Description: as for outcome 6
Time Frame: 42 days after the fourth dose
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 361 | 126
Participants | 358 | 125
Statistical Analysis 1: Comparison: Menhibrix Group vs ActHIB Group; To demonstrate that, following a fourth dose, the immune response to Hib polysaccharide (PRP) in the group that received 3 primary vaccine doses of Menhibrix vaccine and a fourth dose of Menhibrix vaccine coadministered with M-M-R II and Varivax vaccines was non-inferior to the corresponding immune response in the group that received 3 primary vaccine doses of ActHIB vaccine and a fourth dose of PedvaxHIB vaccine co-administered with M-M-R II and Varivax vaccines; Test type: Non-Inferiority — Criteria for non-inferiority (42 days after the fourth dose): Lower limit of the two-sided standardized asymptotic 95% CI on the difference (Menhibrix vaccine fourth dose group minus ActHIB fourth dose group) in the percentage of subjects with anti-PRP concentration ≥ 1.0 µg/mL is ≥ -10% (clinical limit for non-inferiority); Difference in percentage = -0.04, 95% CI 2-sided [-1.78 to 3.57]

11. Primary Outcome: Number of Subjects With Anti-mumps Titer Equal to or Above 28 Estimated Dose 50 (ED50)
Description: The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-mumps antibody titers below 28 ED50
  Co-administration with MMR-II vaccine.
Time Frame: 42 days after the fourth dose
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 601 | 191
Participants | 595 | 191
Statistical Analysis 1: Comparison: Menhibrix Group vs ActHIB Group; To demonstrate the non-inferiority of M-M-R II vaccine when co-administered with a fourth dose of Menhibrix vaccine compared to M--M-R II vaccine co-administered with a fourth dose of PedvaxHIB vaccine, each co-administered with Varivax vaccine; Test type: Non-Inferiority — Criterion for non-inferiority (42 days after fourth dose vaccination): Lower limit of the standardized asymptotic 95% CI for the difference (Menhibrix vaccine fourth dose group minus ActHIB fourth dose group) in the percentage of subjects with a seroconversion ≥28 ED50, in subjects with initial anti-mumps antibody < 28 ED50, for anti-mumps antibody is ≥ -5% (clinical limit for non-inferiority); Difference in percentage = -1, 95% CI 2-sided [-2.16 to 0.98]

12. Primary Outcome: Number of Subjects With Anti-rubella Antibody Concentrations Equal to or Above 10 International Units Per Milli-litre (IU/mL)
Description: The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-measles antibody concentrations below 4 IU/mL.
  Co-administration with MMR-II vaccine.
Time Frame: 42 days after the fourth dose
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 850 | 285
Participants | 848 | 284
Statistical Analysis 1: Comparison: Menhibrix Group vs ActHIB Group; [analysis description as in outcome 9, analysis 1]; Test type: Non-Inferiority — Criterion for non-inferiority (42 days after fourth dose vaccination): Lower limit of the standardized asymptotic 95% CI for the difference (Menhibrix vaccine fourth dose group minus ActHIB fourth dose group) in the percentage of subjects with seroresponse ≥10 IU/ml, in initially seronegative subjects (< 4 IU/ml), for anti-rubella antibody is ≥ -5% (clinical limit for non-inferiority); Difference in percentage = 0.12, 95% CI 2-sided [-0.57 to 1.73]

13. Primary Outcome: Number of Subjects With Anti-varicella Titer Equal to or Above 1:5
Description: The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-measles antibody titer below 1:5.
  Co-administration with Varivax vaccine.
Time Frame: 42 days after the fourth dose
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 723 | 223
Participants | 722 | 223
Statistical Analysis 1: Comparison: Menhibrix Group vs ActHIB Group; To demonstrate the non-inferiority of Varivax vaccine co-administered with a fourth dose of Menhibrix vaccine compared to Varivax vaccine co-administered with a fourth dose of PedvaxHIB vaccine, each co-administered with M-M-R II vaccine in terms of immunogenicity to varicella as measured by fluorescent antibody to membrane antigen (FAMA); Test type: Non-Inferiority — Criterion for non-inferiority (42 days after the fourth dose vaccination): Lower limit of the standardized asymptotic 95% CI for the difference (Menhibrix vaccine fourth dose group minus ActHIB fourth dose group) in the percentage of subjects with seroconversion ≥ 1:5 dilution, in initially seronegative subjects (< 1:5), for anti-varicella antibody is ≥ -10% (clinical limit for non-inferiority); Difference in percentage = -0.14, 95% CI 2-sided [-0.78 to 1.56]

14. Secondary Outcome: Number of Subjects With Anti-tetanus (Anti-T) and Anti-diphtheria Toxoid (Anti-D) Antibody Concentrations Equal to or Above 0.1 International Units Per Millilitre (IU/mL)
Description: as for outcome 6
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 365 | 120
Participants
  Anti-D | 365 | 120
  Anti-T | 365 | 120

15. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in international units per milliliter (IU/mL).
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 365 | 120
IU/mL
  Anti-D | 2.0 [1.9 to 2.2] | 2.2 [2.0 to 2.5]
  Anti-T | 3.9 [3.7 to 4.1] | 1.9 [1.7 to 2.2]

16. Secondary Outcome: Number of Subjects With Anti Hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Equal to or Above 10.0 Milli-international Units Per Millilitre (mIU/mL)
Description: Results are stratified by the presence or absence of a birth dose of hepatitis B vaccine.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 194 | 47
Participants
  Anti-HBs with Hepatitis B at birth | 193 | 47
  Anti-HBs without Hepatitis B at birth: number analyzed (Participants) | 18 | 8
  Anti-HBs without Hepatitis B at birth | 17 | 8

17. Secondary Outcome: Anti-HBS Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in milli-International units per milliliter (mIU/mL)
  Results are stratified by the presence or absence of a birth dose of hepatitis B vaccine.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 194 | 47
mIU/mL
  Anti-HBs with Hepatitis B at birth | 1963.2 [1684.8 to 2287.7] | 2187.6 [1551.4 to 3084.5]
  Anti-HBs without Hepatitis B at birth: number analyzed (Participants) | 18 | 8
  Anti-HBs without Hepatitis B at birth | 1672.7 [730.9 to 3827.8] | 3593.2 [1499.4 to 8611.1]

18. Secondary Outcome: Number of Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations Equal to or Above 5 ELISA Units Per Millilitre (EL.U/mL)
Description: as for outcome 6
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 327 | 101
Participants
  Anti-PT: number analyzed (Participants) | 327 | 100
  Anti-PT | 327 | 100
  Anti-FHA: number analyzed (Participants) | 324 | 97
  Anti-FHA | 324 | 97
  Anti-PRN: number analyzed (Participants) | 322 | 101
  Anti-PRN | 321 | 99

19. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: as for outcome 6
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 327 | 101
EL.U/mL
  Anti-PT: number analyzed (Participants) | 327 | 100
  Anti-PT | 57.7 [54.0 to 61.7] | 65.6 [58.3 to 73.9]
  Anti-FHA: number analyzed (Participants) | 324 | 97
  Anti-FHA | 243.8 [227.9 to 260.9] | 293.6 [261.4 to 329.8]
  Anti-PRN: number analyzed (Participants) | 322 | 101
  Anti-PRN | 98.6 [89.5 to 108.6] | 103.1 [82.8 to 128.4]

20. Secondary Outcome: Number of Subjects With Anti-poliovirus Types 1, 2 and 3 Equal to or Above 8 Estimated Dose 50 (ED50)
Description: as for outcome 6
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 285 | 90
Participants
  Anti-Polio 1 | 285 | 90
  Anti-Polio 2 | 285 | 90
  Anti-Polio 3: number analyzed (Participants) | 285 | 89
  Anti-Polio 3 | 285 | 89

21. Secondary Outcome: Anti-poliovirus Types 1, 2 and 3 Titers
Description: as for outcome 4
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 285 | 90
Titers
  Anti-Polio 1 | 591.8 [525.0 to 667.0] | 590.7 [462.7 to 754.1]
  Anti-Polio 2 | 496.7 [435.9 to 566.0] | 452.7 [360.3 to 568.8]
  Anti-Polio 3: number analyzed (Participants) | 285 | 89
  Anti-Polio 3 | 1367.7 [1209.9 to 1546.0] | 1239.2 [973.5 to 1577.6]

22. Secondary Outcome: Number of Subjects With Antibodies to Neisseria Meningitidis Serogroup C and Y Polysaccharide Capsule (Anti-PSC and Anti-PSY) Concentrations Equal to or Above the Cut-off Values
Description: Anti-PSC and anti-PSY antibody cut-off values assessed were >=0.3 microgram per milliliter (µg/mL) and >=2.0 µg/mL.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 421 | 119
Participants
  Anti-PSC >=0.3 µg/mL | 418 | 5
  Anti-PSY >=0.3 µg/mL: number analyzed (Participants) | 404 | 109
  Anti-PSY >=0.3 µg/mL | 402 | 1
  Anti-PSC >=2.0 µg/mL | 379 | 2
  Anti-PSY >=2.0 µg/mL: number analyzed (Participants) | 404 | 109
  Anti-PSY >=2.0 µg/mL | 396 | 0

23. Secondary Outcome: Anti-PSC and Anti-PSY Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in microgram per milliliter (µg/mL)
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 421 | 119
µg/mL
  Anti-PSC | 5.8 [5.3 to 6.2] | 0.2 [0.2 to 0.2]
  Anti-PSY: number analyzed (Participants) | 404 | 109
  Anti-PSY | 17.5 [16.0 to 19.1] | 0.2 [0.1 to 0.2]

24. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations Equal to or Above the Cut-off Values
Description: Anti-PRP antibody cut-off values assessed were >=0.15 microgram per milliliter (µg/mL) and >=1.0 µg/mL.
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: One month after the primary vaccination course
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 49 | 42 | 43 | 134 | 46
Participants
  Anti-PRP >=0.15 µg/mL | 49 | 42 | 43 | 134 | 46
  Anti-PRP >=1.0 µg/mL | 49 | 42 | 43 | 134 | 46

25. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations Equal to or Above the Cut-off Values
Description: as for outcome 24
Time Frame: Prior to the fourth dose vaccination and one month after fourth dose vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 40 | 13
Participants
  Anti-PRP pre-dose 4 >=0.15 µg/mL: number analyzed (Participants) | 38 | 12
  Anti-PRP pre-dose 4 >=0.15 µg/mL | 38 | 12
  Anti-PRP pre-dose 4 >=1.0 µg/mL: number analyzed (Participants) | 38 | 12
  Anti-PRP pre-dose 4 >=1.0 µg/mL | 33 | 11
  Anti-PRP post-dose 4 >=0.15 µg/mL | 40 | 13
  Anti-PRP post-dose 4 >=1.0 µg/mL | 40 | 13

26. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in microgram per millilitre (µg/mL)
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: One month after the primary vaccination course
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 49 | 42 | 43 | 134 | 46
µg/mL | 24.984 [19.674 to 31.728] | 24.050 [18.327 to 31.561] | 20.489 [15.653 to 26.819] | 23.165 [20.012 to 26.815] | 29.759 [22.729 to 38.965]

27. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: as for outcome 26
Time Frame: Prior to the fourth dose vaccination and one month after fourth dose vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 40 | 13
µg/mL
  Anti-PRP Pre-dose 4: number analyzed (Participants) | 38 | 12
  Anti-PRP Pre-dose 4 | 3.340 [2.407 to 4.636] | 4.123 [1.981 to 8.583]
  Anti-PRP Post-dose 4 | 132.965 [97.131 to 182.019] | 92.800 [45.636 to 188.709]

28. Secondary Outcome: Number of Subjects With hSBA-MenC and hSBA-MenY Titers Equal to or Above the Cut-off Values
Description: hSBA-MenC/Y antibody cut-off values assessed were >=1:4 and >=1:8
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: One month after the primary vaccination course
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 49 | 42 | 44 | 135 | 46
Participants
  hSBA-MenC >=1:4: number analyzed (Participants) | 48 | 42 | 44 | 134 | 46
  hSBA-MenC >=1:4 | 47 | 42 | 44 | 133 | 2
  hSBA-MenC >=1:8: number analyzed (Participants) | 48 | 42 | 44 | 134 | 46
  hSBA-MenC >=1:8 | 47 | 42 | 44 | 133 | 2
  hSBA-MenY >=1:4: number analyzed (Participants) | 49 | 42 | 44 | 135 | 45
  hSBA-MenY >=1:4 | 48 | 42 | 44 | 134 | 1
  hSBA-MenY >=1:8: number analyzed (Participants) | 49 | 42 | 44 | 135 | 45
  hSBA-MenY >=1:8 | 48 | 42 | 44 | 134 | 1

29. Secondary Outcome: Number of Subjects With hSBA-MenC and hSBA-MenY Titers Equal to or Above the Cut-off Values
Description: hSBA-MenC/Y antibody cut-off values assessed were >=1:4 and >=1:8.
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: Prior to the fourth dose vaccination and one month after fourth dose vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 40 | 13
Participants
  hSBA-MenC pre-dose 4 >=1:4: number analyzed (Participants) | 39 | 13
  hSBA-MenC pre-dose 4 >=1:4 | 39 | 2
  hSBA-MenC pre-dose 4 >=1:8: number analyzed (Participants) | 39 | 13
  hSBA-MenC pre-dose 4 >=1:8 | 39 | 2
  hSBA-MenC post-dose 4 >=1:4: number analyzed (Participants) | 39 | 13
  hSBA-MenC post-dose 4 >=1:4 | 39 | 1
  hSBA-MenC post-dose 4 >=1:8: number analyzed (Participants) | 39 | 13
  hSBA-MenC post-dose 4 >=1:8 | 39 | 1
  hSBA-MenY pre-dose 4 >=1:4: number analyzed (Participants) | 39 | 13
  hSBA-MenY pre-dose 4 >=1:4 | 39 | 3
  hSBA-MenY pre-dose 4 >=1:8: number analyzed (Participants) | 39 | 13
  hSBA-MenY pre-dose 4 >=1:8 | 39 | 3
  hSBA-MenY post-dose 4 >=1:4 | 40 | 7
  hSBA-MenY post-dose 4 >=1:8 | 40 | 7

30. Secondary Outcome: hSBA-MenC and hSBA-MenY Antibody Titers
Description: Titres are expressed as Geometric Mean Titers (GMTs).
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: One month after the primary vaccination course
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 49 | 42 | 44 | 135 | 46
Titers
  hSBA-MenC: number analyzed (Participants) | 48 | 42 | 44 | 134 | 46
  hSBA-MenC | 3055.8 [2096.8 to 4453.6] | 3370.7 [2545.4 to 4463.6] | 3119.3 [2418.9 to 4022.4] | 3172.6 [2657.9 to 3786.8] | 2.4 [1.8 to 3.1]
  hSBA-MenY: number analyzed (Participants) | 49 | 42 | 44 | 135 | 45
  hSBA-MenY | 666.5 [464.0 to 957.3] | 916.7 [666.9 to 1260.1] | 989.6 [756.7 to 1294.2] | 837.2 [696.4 to 1006.3] | 2.2 [1.8 to 2.5]

31. Secondary Outcome: hSBA-MenC and hSBA-MenY Antibody Titers
Description: Titers are expressed as Geometric Mean Titers (GMTs)
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: Prior to the fourth dose vaccination and one month after fourth dose vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 40 | 13
Titers
  hSBA-MenC pre-dose 4: number analyzed (Participants) | 39 | 13
  hSBA-MenC pre-dose 4 | 504.7 [366.2 to 695.5] | 3.6 [1.5 to 8.7]
  hSBA-MenC post-dose 4: number analyzed (Participants) | 39 | 13
  hSBA-MenC post-dose 4 | 10132.9 [8008.0 to 12821.7] | 2.5 [1.6 to 3.8]
  hSBA-MenY pre-dose 4: number analyzed (Participants) | 39 | 13
  hSBA-MenY pre-dose 4 | 446.5 [328.3 to 607.3] | 5.3 [1.7 to 16.7]
  hSBA-MenY post-dose 4 | 5775.8 [4488.9 to 7431.7] | 27.4 [5.8 to 129.0]

32. Secondary Outcome: Number of Subjects With Anti-PSC and Anti-PSY Antibody Concentrations Equal to or Above the Cut-off Values
Description: Anti-PSC and anti-PSY antibody cut-off values assessed were >=0.3 microgram per milliliter (µg/mL) and >=2.0 µg/mL.
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: One month after the primary vaccination course
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 134 | 46
Participants
  Anti-PSC >=0.3 µg/mL | 134 | 2
  Anti-PSC >=2.0 µg/mL | 134 | 1
  Anti-PSY >=0.3 µg/mL: number analyzed (Participants) | 130 | 46
  Anti-PSY >=0.3 µg/mL | 130 | 1
  Anti-PSY >=2.0 µg/mL: number analyzed (Participants) | 130 | 46
  Anti-PSY >=2.0 µg/mL | 130 | 1

33. Secondary Outcome: Number of Subjects With Anti-PSC and Anti-PSY Antibody Concentrations Equal to or Above the Cut-off Values
Description: Anti-PSC and anti-PSY antibody cut-off values assessed were >=0.3 µg/mL and >=2.0 µg/mL.
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: Prior to the fourth dose vaccination and one month after fourth dose vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 40 | 13
Participants
  Anti-PSC pre-dose 4 >=0.3 µg/mL | 40 | 0
  Anti-PSC pre-dose 4 >=2.0 µg/mL | 22 | 0
  Anti-PSC post-dose 4 >=0.3 µg/mL: number analyzed (Participants) | 39 | 13
  Anti-PSC post-dose 4 >=0.3 µg/mL | 39 | 0
  Anti-PSC post-dose 4 >=2.0 µg/mL: number analyzed (Participants) | 39 | 13
  Anti-PSC post-dose 4 >=2.0 µg/mL | 39 | 0
  Anti-PSY pre-dose 4 >=0.3 µg/mL | 40 | 0
  Anti-PSY pre-dose 4 >=2.0 µg/mL | 36 | 0
  Anti-PSY post-dose 4 >=0.3 µg/mL | 40 | 0
  Anti-PSY post-dose 4 >=2.0 µg/mL | 40 | 0

34. Secondary Outcome: Anti-PSC and Anti-PSY Antibodies Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in microgram per milliliter (µg/mL).
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: One month after the primary vaccination course
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 134 | 46
µg/mL
  Anti-PSC | 13.4 [12.1 to 15.0] | 0.2 [0.1 to 0.2]
  Anti-PSY: number analyzed (Participants) | 130 | 46
  Anti-PSY | 36.7 [32.2 to 41.8] | 0.2 [0.1 to 0.2]

35. Secondary Outcome: Anti-PSC and Anti-PSY Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in microgram per millilitre (µg/mL).
  The analysis was performed on the cohort 3 (Non-US Safety and Immunogenicity): Cohort 3 was to include the subjects enrolled at 1 center in Mexico. Only descriptive immunogenicity results were reported for this cohort. These subjects also contributed to the safety analysis.
Time Frame: Prior to the fourth dose vaccination and one month after fourth dose vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 40 | 13
µg/mL
  Anti-PSC pre-dose 4 | 2.20 [1.72 to 2.83] | 0.15 [0.15 to 0.15]
  Anti-PSC post-dose 4: number analyzed (Participants) | 39 | 13
  Anti-PSC post-dose 4 | 15.63 [13.30 to 18.37] | 0.15 [0.15 to 0.15]
  Anti-PSY pre-dose 4 | 5.70 [4.18 to 7.78] | 0.15 [0.15 to 0.15]
  Anti-PSY post-dose 4 | 64.66 [52.35 to 79.86] | 0.15 [0.15 to 0.15]

36. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations Equal to or Above the Cut-off Value
Description: Anti-PRP antibody cut-off values assessed were >=0.15 µg/mL.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after the primary vaccination course
Population: The Primary ATP cohort for immunogenicity included evaluable subjects (i.e. those who met eligibility criteria, complied with the procedures and met no elimination criteria) for whom assay results were available for antibodies against at least 1 study vaccine antigen for the blood sample taken during primary vaccination (after the 3rd vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group
Number analyzed (Participants) | 518 | 171 | 162 | 180 | 176
Participants | 518 | 168 | 162 | 180 | 176

37. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in microgram per millilitre (µg/mL).
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after the primary vaccination course and prior to the fourth dose vaccination
Population: The Fourth dose ATP cohort for safety included eligible subjects, who met inclusion criteria, who received 3 vaccine doses in the primary vaccination course, who received the fourth vaccine dose, who did not receive a vaccine not specified or forbidden and who were not excluded from from the Primary ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 469 | 160
µg/mL
  Anti-PRP post-primary | 10.802 [9.767 to 11.947] | 6.086 [4.897 to 7.564]
  Anti-PRP pre-dose 4: number analyzed (Participants) | 441 | 147
  Anti-PRP pre-dose 4 | 1.615 [1.439 to 1.812] | 0.832 [0.664 to 1.042]

38. Secondary Outcome: Number of Subjects With hSBA-MenC and hSBA-MenY Antibody Titers Equal to or Above the Cut-off Values
Description: hSBA-MenC and hSBA-MenY antibody cut-off values assessed were >=1:4 and >=1:8.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: One month after the primary vaccination course
Population: The Primary ATP cohort for immunogenicity included evaluable subjects (i.e. those who met eligibility criteria, complied with the procedures and met no elimination criteria ) for whom assay results were available for antibodies against at least 1 study vaccine antigen for the blood sample taken during primary vaccination (after the 3rd vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group | Menhibrix A Group | Menhibrix B Group | Menhibrix C Group
Number analyzed (Participants) | 491 | 164 | 158 | 168 | 165
Participants
  hSBA-MenC >=1:4 | 485 | 11 | 156 | 167 | 162
  hSBA-MenC >=1:8 | 485 | 11 | 156 | 167 | 162
  hSBA-MenY >=1:4: number analyzed (Participants) | 481 | 162 | 150 | 168 | 163
  hSBA-MenY >=1:4 | 463 | 3 | 141 | 165 | 157
  hSBA-MenY >=1:8: number analyzed (Participants) | 481 | 162 | 150 | 168 | 163
  hSBA-MenY >=1:8 | 461 | 3 | 140 | 165 | 156

39. Secondary Outcome: Number of Subjects With Anti-PSC and Anti-PSY Antibody Concentrations Equal to or Above the Cut-off Values
Description: Anti-PSC and anti-PSY antibody cut-off values assessed were >=0.3 µg/mL and >=2.0 µg/mL.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: Prior to the fourth dose vaccination and 42 days after fourth dose vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 334 | 109
Participants
  Anti-PSC pre-dose 4 >=0.3 µg/mL: number analyzed (Participants) | 327 | 99
  Anti-PSC pre-dose 4 >=0.3 µg/mL | 300 | 3
  Anti-PSC pre-dose 4 >=2.0 µg/mL: number analyzed (Participants) | 327 | 99
  Anti-PSC pre-dose 4 >=2.0 µg/mL | 73 | 0
  Anti-PSC post-dose 4 >=0.3 µg/mL: number analyzed (Participants) | 316 | 106
  Anti-PSC post-dose 4 >=0.3 µg/mL | 313 | 9
  Anti-PSC post-dose 4 >=2.0 µg/mL: number analyzed (Participants) | 316 | 106
  Anti-PSC post-dose 4 >=2.0 µg/mL | 262 | 6
  Anti-PSY pre-dose 4 >=0.3 µg/mL: number analyzed (Participants) | 325 | 93
  Anti-PSY pre-dose 4 >=0.3 µg/mL | 320 | 1
  Anti-PSY pre-dose 4 >=2.0 µg/mL: number analyzed (Participants) | 325 | 93
  Anti-PSY pre-dose 4 >=2.0 µg/mL | 235 | 0
  Anti-PSY post-dose 4 >=0.3 µg/mL | 332 | 6
  Anti-PSY post-dose 4 >=2.0 µg/mL | 325 | 4

40. Secondary Outcome: Anti-PSC and Anti-PSY Antibody Concentrations
Description: as for outcome 37
Time Frame: Prior to the fourth dose vaccination and 42 days after fourth dose vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 334 | 109
µg/mL
  Anti-PSC pre-dose 4: number analyzed (Participants) | 327 | 99
  Anti-PSC pre-dose 4 | 1.04 [0.94 to 1.16] | 0.16 [0.15 to 0.17]
  Anti-PSC post-dose 4: number analyzed (Participants) | 316 | 106
  Anti-PSC post-dose 4 | 4.81 [4.33 to 5.34] | 0.19 [0.16 to 0.23]
  Anti-PSY pre-dose 4: number analyzed (Participants) | 325 | 93
  Anti-PSY pre-dose 4 | 3.15 [2.83 to 3.50] | 0.15 [0.15 to 0.15]
  Anti-PSY post-dose 4 | 18.26 [16.41 to 20.31] | 0.18 [0.15 to 0.21]

41. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations Equal to or Above 0.15 Microgram Per Milliliter (µg/mL)
Description: as for outcome 6
Time Frame: Prior to the fourth dose vaccination and 42 days after fourth vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 361 | 126
Participants
  Anti-PRP [post-dose 4] | 361 | 126
  Anti-PRP [pre-dose 4]: number analyzed (Participants) | 341 | 112
  Anti-PRP [pre-dose 4] | 329 | 98

42. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: as for outcome 1
Time Frame: Prior to the fourth vaccination and 42 days after fourth vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 361 | 126
µg/mL
  Anti-PRP [post-dose 4] | 34.851 [30.664 to 39.610] | 20.200 [16.373 to 24.920]
  Anti-PRP [pre-dose 4]: number analyzed (Participants) | 341 | 112
  Anti-PRP [pre-dose 4] | 1.617 [1.420 to 1.842] | 0.759 [0.589 to 0.978]

43. Secondary Outcome: Number of Subjects With hSBA-MenC and hSBA-MenY Antibody Concentrations Equal to or Above 1:4
Description: as for outcome 6
Time Frame: Prior to the fourth dose vaccination and 42 days after fourth vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 342 | 120
Participants
  hSBA-MenC [post-dose 4]: number analyzed (Participants) | 331 | 119
  hSBA-MenC [post-dose 4] | 326 | 26
  hSBA-MenY [post-dose 4] | 338 | 87
  hSBA-MenC [pre-dose 4]: number analyzed (Participants) | 329 | 104
  hSBA-MenC [pre-dose 4] | 318 | 12
  hSBA-MenY [pre-dose 4]: number analyzed (Participants) | 329 | 103
  hSBA-MenY [pre-dose 4] | 309 | 6

44. Secondary Outcome: Number of Subjects With Anti-measles Antibody Concentrations Equal to or Above 200 Milli-international Units Per Millilitre (mIU/mL)
Description: The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-measles antibody concentrations below 150 mIU/mL.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: 42 days after fourth vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 852 | 286
Participants | 812 | 273

45. Secondary Outcome: Anti-measles Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in milli-international units per milliliter (mIU/mL).
  The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-measles antibody concentrations below 150 mIU/mL.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: 42 days after fourth vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 852 | 286
mIU/mL | 1990.0 [1852.2 to 2138.0] | 1989.5 [1765.4 to 2242.2]

46. Secondary Outcome: Number of Subjects With Anti-mumps Titer Equal to or Above the Cut-off Values
Description: Anti-mumps antibody cut-off values assessed were >=28 estimated dose 50 (ED50) and >=51 ED50.
  The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-mumps antibody titers below 24 ED50.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: 42 days after fourth vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 536 | 176
Participants
  Anti-mumps >=28 ED50 | 532 | 176
  Anti-mumps >=51 ED50 | 490 | 160

47. Secondary Outcome: Anti-mumps Antibody Titers
Description: Titers are expressed as Geometric Mean Titers (GMTs).
  The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-measles antibody titers below 24 ED50.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: 42 days after fourth vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 536 | 176
Titers | 123.9 [116.9 to 131.3] | 114.3 [103.7 to 126.0]

48. Secondary Outcome: Number of Subjects With Anti-rubella Antibody Concentrations Equal to or Above 4 International Units Per Millilitre (IU/mL)
Description: The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-rubella antibody concentrations below 4 IU/mL.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: 42 days after fourth vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 850 | 285
Participants | 850 | 285

49. Secondary Outcome: Anti-rubella Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) and are expressed in international units per milliliter (IU/mL).
  The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-rubella antibody concentrations below 4 IU/mL.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: 42 days after fourth vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 850 | 285
IU/mL | 81.4 [77.5 to 85.4] | 74.9 [68.9 to 81.4]

50. Secondary Outcome: Number of Subjects With Anti-varicella Titer Equal to or Above 1:40
Description: The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-rubella antibody concentrations below 1:5
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: 42 days after fourth vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 723 | 223
Participants | 722 | 223

51. Secondary Outcome: Anti-varicella Antibody Titers
Description: Titers are expressed as Geometric Mean Titers (GMTs)
  The analysis was performed on initially seronegative subjects. Seronegative subjects are subjects with anti-varicella antibody titers below 1:5
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based. These subjects also contributed to the safety analysis.
Time Frame: 42 days after fourth vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 723 | 223
Titers | 407.1 [389.4 to 425.5] | 394.1 [364.6 to 426.0]

52. Secondary Outcome: Number of Subjects With Anti-H1N1, Anti-H3N2 and Anti-influenza-B (Anti B) Antibody Titers Equal to or Above 1:40
Description: anti-H1N1, anti-H3N2 and anti-influenza-B (anti B) antibody were measured by hemagglutination inhibition assay (HIA), in subjects who received 2 doses of influenza vaccine within the same influenza season of which at least one dose is concomitant with the study vaccine. For the purposes of this study, concomitant administration of influenza vaccine was defined as administration within 28 days before to 7 days after administration of study vaccines.
  This analysis occurred on the cohort 1: Cohort 1 was to include subjects in the US on which all immunogenicity analyses were to be based.
Time Frame: Prior to the fourth dose vaccination and one month after the fourth dose vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 5 | 4
Participants
  Anti-H1N1 pre-dose 4: number analyzed (Participants) | 5 | 3
  Anti-H1N1 pre-dose 4 | 0 | 0
  Anti-H1N1 post-dose 4: number analyzed (Participants) | 4 | 4
  Anti-H1N1 post-dose 4 | 2 | 1
  Anti-H3N2 pre-dose 4: number analyzed (Participants) | 5 | 3
  Anti-H3N2 pre-dose 4 | 0 | 0
  Anti-H3N2 post-dose 4: number analyzed (Participants) | 4 | 4
  Anti-H3N2 post-dose 4 | 3 | 1
  Anti-B pre-dose 4: number analyzed (Participants) | 5 | 3
  Anti-B pre-dose 4 | 0 | 0
  Anti-B post-dose 4: number analyzed (Participants) | 4 | 4
  Anti-B post-dose 4 | 1 | 1

53. Secondary Outcome: Number of Subjects Reporting Fever Above 39.5 Degrees Celsius/103.1 Degrees Fahrenheit
Description: Fever is defined as temperature (rectal or axillary/tympanic) above 39.5 degrees Celsius (°C) or 103.1 degrees Fahrenheit (°F).
Time Frame: In the 4-day (Day 0-3) follow-up period after primary vaccination course
Population: The Primary Total Vaccinated cohort included all vaccinated subjects (Cohort 1, Cohort 2 & Cohort 3) in the primary phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3089 | 1015
Participants | 46 | 16

54. Secondary Outcome: Number of Subjects Reporting Fever Above 39.5 Degrees Celsius/103.1 Degrees Fahrenheit
Description: as for outcome 53
Time Frame: In the 4-day (Day0-3) follow-up period after the fourth dose
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 2527 | 831
Participants | 18 | 5

55. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Solicited genral symptoms assessed were fever, irritability/fussiness, drowsiness and loss of appetite. Fever is defined as temperature (rectal or axillary/tympanic) equal to or above 38.0°C.
Time Frame: Within the 4 days (Day 0-3) following each dose of the primary vaccination course
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3089 | 1016
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 3056 | 1008
  Any Pain, Dose 1 | 1849 | 672
  Any Pain, Dose 2: number analyzed (Participants) | 2903 | 954
  Any Pain, Dose 2 | 1679 | 596
  Any Pain, Dose 3: number analyzed (Participants) | 2740 | 904
  Any Pain, Dose 3 | 1454 | 522
  Any Pain, Across doses: number analyzed (Participants) | 3088 | 1016
  Any Pain, Across doses | 2419 | 819
  Any Redness, Dose 1: number analyzed (Participants) | 3056 | 1008
  Any Redness, Dose 1 | 1152 | 401
  Any Redness, Dose 2: number analyzed (Participants) | 2903 | 954
  Any Redness, Dose 2 | 1455 | 483
  Any Redness, Dose 3: number analyzed (Participants) | 2740 | 904
  Any Redness, Dose 3 | 1409 | 495
  Any Redness, Across doses: number analyzed (Participants) | 3088 | 1016
  Any Redness, Across doses | 2052 | 691
  Any Swelling, Dose 1: number analyzed (Participants) | 3056 | 1008
  Any Swelling, Dose 1 | 893 | 281
  Any Swelling, Dose 2: number analyzed (Participants) | 2903 | 954
  Any Swelling, Dose 2 | 1091 | 350
  Any Swelling, Dose 3: number analyzed (Participants) | 2740 | 904
  Any Swelling, Dose 3 | 1110 | 381
  Any Swelling, Across doses: number analyzed (Participants) | 3088 | 1016
  Any Swelling, Across doses | 1707 | 568
  Any Drowsiness, Dose 1: number analyzed (Participants) | 3055 | 1008
  Any Drowsiness, Dose 1 | 1864 | 655
  Any Drowsiness, Dose 2: number analyzed (Participants) | 2900 | 952
  Any Drowsiness, Dose 2 | 1588 | 552
  Any Drowsiness, Dose 3: number analyzed (Participants) | 2736 | 905
  Any Drowsiness, Dose 3 | 1260 | 444
  Any Drowsiness, Across doses: number analyzed (Participants) | 3088 | 1015
  Any Drowsiness, Across doses | 2418 | 804
  Any Temperature, Dose 1: number analyzed (Participants) | 3056 | 1008
  Any Temperature, Dose 1 | 688 | 228
  Any Temperature, Dose 2: number analyzed (Participants) | 2900 | 951
  Any Temperature, Dose 2 | 803 | 276
  Any Temperature, Dose 3: number analyzed (Participants) | 2736 | 905
  Any Temperature, Dose 3 | 609 | 206
  Any Temperature, Across doses: number analyzed (Participants) | 3089 | 1015
  Any Temperature, Across doses | 1434 | 463
  Any Irritability, Dose 1: number analyzed (Participants) | 3055 | 1008
  Any Irritability, Dose 1 | 2156 | 782
  Any Irritability, Dose 2: number analyzed (Participants) | 2900 | 952
  Any Irritability, Dose 2 | 2074 | 708
  Any Irritability, Dose 3: number analyzed (Participants) | 2736 | 905
  Any Irritability, Dose 3 | 1771 | 600
  Any Irritability, Across doses: number analyzed (Participants) | 3088 | 1015
  Any Irritability, Across doses | 2740 | 926
  Any Loss of appetite, Dose 1: number analyzed (Participants) | 3055 | 1008
  Any Loss of appetite, Dose 1 | 1024 | 375
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 2900 | 952
  Any Loss of appetite, Dose 2 | 921 | 317
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 2736 | 905
  Any Loss of appetite, Dose 3 | 828 | 285
  Any Loss of appetite, Across doses: number analyzed (Participants) | 3088 | 1015
  Any Loss of appetite, Across doses | 1764 | 609

56. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms assessed were pain, redness, swelling and an increase in limb circumference. Solicited general symptoms assessed were fever, irritability/fussiness, drowsiness and lost of appetite. Fever is defined as temperature (rectal or axillary/tympanic) equal to or above 38.0°C
Time Frame: Within the 4 days (Day 0-3) post-vaccination period following the fourth dose
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 2769 | 923
Participants
  Pain: number analyzed (Participants) | 2528 | 832
  Pain | 1319 | 494
  Redness: number analyzed (Participants) | 2528 | 833
  Redness | 1213 | 463
  Swelling: number analyzed (Participants) | 2526 | 832
  Swelling | 936 | 334
  Increase in limb circumference | 1489 | 503
  Drowsiness: number analyzed (Participants) | 2526 | 830
  Drowsiness | 1088 | 381
  Fever: number analyzed (Participants) | 2527 | 831
  Fever | 341 | 134
  Irritability: number analyzed (Participants) | 2526 | 830
  Irritability | 1482 | 534
  Loss of appetite: number analyzed (Participants) | 2526 | 830
  Loss of appetite | 825 | 287

57. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 31 days (Day 0-30) following the primary vaccination course
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3136 | 1044
Participants | 1820 | 602

58. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: as for outcome 57
Time Frame: Within 31 days (Day 0-30) following the fourth dose
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 2769 | 923
Participants | 1010 | 334

59. Secondary Outcome: Number of Subjects Reporting Increased Circumferential Swelling at the Injection Limb(s)
Description: Increased circumferential swelling defined as either swelling with a diameter of >50 mm or a >50 mm increase in the circumference of the mid-limb when compared to the baseline (pre-vaccination) measurement, or any diffuse swelling that interferes with or prevents everyday activities (for example, active playing, eating, sleeping).
Time Frame: Within 4 days (Day 0 to Day 3) after fourth dose vaccination
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 2769 | 923
Participants | 1489 | 503

60. Secondary Outcome: Number of Subjects Reporting General Symptoms Specific to Measles, Mumps, Rubella and Varicella Vaccination
Description: Symptoms assessed were fever, rash/exanthem, parotid/salivary gland swelling, and any suspected signs of meningism including febrile convulsions. Fever is defined as temperature (rectal or axillary/tympanic) equal to or above 38.0°C.
Time Frame: Within 43 days (Day 0 through Day 42) after vaccination
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 545 | 175
Participants
  Meningismus: number analyzed (Participants) | 541 | 173
  Meningismus | 0 | 0
  Parotiditis: number analyzed (Participants) | 541 | 173
  Parotiditis | 0 | 0
  Rash: number analyzed (Participants) | 544 | 175
  Rash | 59 | 19
  Fever: number analyzed (Participants) | 545 | 173
  Fever | 211 | 70

61. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: From Dose 0 through 6 months after the last primary dose or untill administration of the fourth dose
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3136 | 1044
Participants | 126 | 50

62. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: as for outcome 61
Time Frame: From the fourth dose through the end of the 6-month safety follow-up
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 2769 | 923
Participants | 47 | 18

63. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Illness(es) (NOCDs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From Dose 0 through 6 months after the last primary dose or until administration of the fourth dose
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3136 | 1044
Participants | 163 | 52

64. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Illness(es) (NOCDs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From the fourth dose through the end of the 6-month safety follow-up
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 2769 | 923
Participants | 85 | 33

65. Secondary Outcome: Number of Subjects Reporting Rash
Description: Rash assessed was hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: From Dose 0 through 6 months after the last primary dose or until administration of the fourth dose
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3136 | 1044
Participants | 470 | 154

66. Secondary Outcome: Number of Subjects Reporting Rash
Description: Rash assessed was hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: From the fourth dose through the end of the 6-month safety follow-up
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 2769 | 923
Participants | 265 | 94

67. Secondary Outcome: Number of Subjects Reporting Adverse Events Resulting in Emergency Room (ER) Visits
Description: Emergency room (ER) visits were not related to well-child care, vaccination, injury or common acute illness such as upper respiratory tract infections; otitis media, pharyngitis, gastroenteritis.
Time Frame: From Dose 0 through 6 months after the last primary dose or until administration of the fourth dose
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3136 | 1044
Participants | 217 | 72

68. Secondary Outcome: Number of Subjects Reporting Adverse Events Resulting in Physicians (MD) Office Visits.
Description: Physicians (MD) office visits were not related to well-child care, vaccination, injury or common acute illness such as upper respiratory tract infections; otitis media, pharyngitis, gastroenteritis.
Time Frame: From Dose 0 through 6 months after the last primary dose or until administration of the fourth dose
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 3136 | 1044
Participants | 1336 | 433

69. Secondary Outcome: Number of Subjects Reporting Adverse Events Resulting in Emergency Room (ER) Visits
Description: as for outcome 67
Time Frame: From the fourth dose through the end of the 6-month safety follow-up
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 2769 | 923
Participants | 137 | 54

70. Secondary Outcome: Number of Subjects Reporting Adverse Events Resulting in Physicians (MD) Office Visits
Description: as for outcome 68
Time Frame: From the fourth dose through the end of the 6-month safety follow-up
Population: The Fourth dose Total Vaccinated cohort included all vaccinated subjects in the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 2769 | 923
Participants | 668 | 205

71. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentration Equal to or Above 1.0 Microgram Per Milliliter (µg/mL).
Description: as for outcome 6
Time Frame: Prior to the fourth dose vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 341 | 112
Participants | 227 | 52

72. Secondary Outcome: Number of Subjects With hSBA-MenC and hSBA-MenY Antibody Titer Equal to or Above 1:8.
Description: as for outcome 6
Time Frame: Prior to the fourth dose vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB Group
Number analyzed (Participants) | 329 | 104
Participants
  hSBA-MenC [pre-dose 4] | 318 | 12
  hSBA-MenY [pre-dose 4]: number analyzed (Participants) | 329 | 103
  hSBA-MenY [pre-dose 4] | 306 | 6

ADVERSE EVENTS:
Time Frame: SAEs: From Day 0 after Dose 1 through the day preceding the fourth dose; From the fourth dose phase through the end of the safety follow-up; AEs: within the 31-day (Day 0-30) post vaccination period; Solicited AEs: Duting the 4-day post vaccination period
Description: Results are presented for the primary phase and the fourth dose phase.
Arm/Group | Menhibrix Group | ActHIB Group
Serious Adverse Events (participants affected / at risk) | 126/3136 | 50/1044
Other Adverse Events (participants affected / at risk) | 3034/3136 | 998/1044
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Menhibrix Group (N=3136) | ActHIB Group (N=1044)
Gastroenteritis (Infections and infestations) | 19 | 7 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Bronchiolitis (Infections and infestations) | 18 | 5 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Dehydration (Metabolism and nutrition disorders) | 15 | 2 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Otitis media (Infections and infestations) | 8 | 4 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Viral infection (Infections and infestations) | 11 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Gastroenteritis rotavirus (Infections and infestations) | 8 | 2 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Pneumonia (Infections and infestations) | 8 | 2 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Respiratory syncytial virus bronchiolitis (Injury, poisoning and procedural complications) | 8 | 2 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Urinary tract infection (Infections and infestations) | 8 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Respiratory syncytial virus infection (Infections and infestations) | 4 | 4 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Intussusception (Gastrointestinal disorders) | 4 | 2 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Pyrexia (General disorders) | 5 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Croup infectious (Infections and infestations) | 2 | 3 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Bronchopneumonia (Infections and infestations) | 1 | 3 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Febrile convulsion (Nervous system disorders) | 2 | 2 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Upper respiratory tract infection (Infections and infestations) | 4 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Vomiting (Gastrointestinal disorders) | 2 | 2 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Cellulitis (Infections and infestations) | 2 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Convulsion (Nervous system disorders) | 2 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Pneumonia viral (Infections and infestations) | 2 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Pyelonephritis (Infections and infestations) | 1 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Viral skin infection (Infections and infestations) | 2 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Abdominal pain (Gastrointestinal disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Abdominal wall abscess (Infections and infestations) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Abscess (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Acarodermatitis (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Acidosis (Metabolism and nutrition disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Aspiration bronchial (Investigations) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Bronchitis viral (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Cerebellar ataxia (Nervous system disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Child maltreatment syndrome (Injury, poisoning and procedural complications) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Conjunctivitis (Eye disorders) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Dacryostenosis acquired (Eye disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Gastroenteritis adenovirus (Infections and infestations) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Gastroenteritis viral (Infections and infestations) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Group b streptococcus neonatal sepsis (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
HIV infection (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Haematemesis (Gastrointestinal disorders) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Head injury (Injury, poisoning and procedural complications) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Hypersensitivity (Immune system disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Hypertension (Vascular disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Hypotonia (Nervous system disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Infantile spasms (Nervous system disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Influenza (Infections and infestations) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Irritability (General disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Lobar pneumonia (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Meningitis viral (Infections and infestations) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Nasopharyngitis (Infections and infestations) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Pertussis (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Sinusitis (Infections and infestations) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Staphylococcal infection (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Sudden infant death syndrome (General disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Tuberous sclerosis (Congenital, familial and genetic disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Typhoid fever (Infections and infestations) | 0 | 1 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Vulval abscess (Infections and infestations) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — From Day 0 after Dose 1 through the day preceding the fourth dose.
Gastroenteritis (Infections and infestations) | 5/2769 | 4/923 — From the fourth dose through the end of the 6-month safety follow-up
Asthma (Respiratory, thoracic and mediastinal disorders) | 4/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Dehydration (Metabolism and nutrition disorders) | 3/2769 | 2/923 — From the fourth dose through the end of the 6-month safety follow-up
Viral infection (Infections and infestations) | 5/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Croup infectious (Infections and infestations) | 4/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Convulsion (Nervous system disorders) | 2/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Head injury (Injury, poisoning and procedural complications) | 1/2769 | 2/923 — From the fourth dose through the end of the 6-month safety follow-up
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Bronchiolitis (Infections and infestations) | 2/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Otitis media (Infections and infestations) | 1/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Pneumonia viral (Infections and infestations) | 1/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Staphylococcal infection (Infections and infestations) | 2/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Abdominal pain (Gastrointestinal disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Abscess (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Abscess neck (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Accidental drug intake by child (Injury, poisoning and procedural complications) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Accidental exposure (Injury, poisoning and procedural complications) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Adenoviral upper respiratory infection (Infections and infestations) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Burns first degree (Injury, poisoning and procedural complications) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Burns second degree (Injury, poisoning and procedural complications) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Cellulitis (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Cellulitis of male external genital organ (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Febrile convulsion (Nervous system disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Gastroenteritis rotavirus (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Gastroenteritis salmonella (Infections and infestations) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Gastroenteritis viral (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Hypersensitivity (Immune system disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Lobar pneumonia (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Lower respiratory tract infection (Infections and infestations) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Lymph node abscess (Infections and infestations) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Lymphadenitis (Blood and lymphatic system disorders) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Multiple injuries (Injury, poisoning and procedural complications) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Neutropenia (Blood and lymphatic system disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Osteomyelitis (Infections and infestations) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Pneumonia (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Pneumonia bacterial (Infections and infestations) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Rash papular (Skin and subcutaneous tissue disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Respiratory tract infection viral (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Seroma (Injury, poisoning and procedural complications) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Skin laceration (Injury, poisoning and procedural complications) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Thermal burn (Injury, poisoning and procedural complications) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Thrombocytopenia (Blood and lymphatic system disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Upper respiratory tract infection (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Urinary tract infection (Infections and infestations) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Urticaria (Skin and subcutaneous tissue disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Ventricular septal defect (Congenital, familial and genetic disorders) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Viral upper respiratory tract infection (Infections and infestations) | 0/2769 | 1/923 — From the fourth dose through the end of the 6-month safety follow-up
Vomiting (Gastrointestinal disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1/2769 | 0/923 — From the fourth dose through the end of the 6-month safety follow-up
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Menhibrix Group (N=3136) | ActHIB Group (N=1044)
Upper respiratory tract infection (Infections and infestations) | 524 | 173 — Within the 31 days (Day 0-30) after the primary vaccination course.
Otitis media (Infections and infestations) | 335 | 104 — Within the 31 days (Day 0-30) after the primary vaccination course.
Vomiting (Gastrointestinal disorders) | 197 | 65 — Within the 31 days (Day 0-30) after the primary vaccination course.
Pyrexia (General disorders) | 176 | 73 — Within the 31 days (Day 0-30) after the primary vaccination course.
Diarrhoea (Gastrointestinal disorders) | 185 | 57 — Within the 31 days (Day 0-30) after the primary vaccination course.
Teething (Gastrointestinal disorders) | 180 | 55 — Within the 31 days (Day 0-30) after the primary vaccination course.
Cough (Respiratory, thoracic and mediastinal disorders) | 163 | 50 — Within the 31 days (Day 0-30) after the primary vaccination course.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 146 | 53 — Within the 31 days (Day 0-30) after the primary vaccination course.
Pyrexia (General disorders) | 176/2769 | 64/923 — Within the 31 days (Day 0-30) after the fourth dose phase
Upper respiratory tract infection (Infections and infestations) | 152/2769 | 50/923 — Within the 31 days (Day 0-30) after the fourth dose phase
Otitis media (Infections and infestations) | 135/2769 | 47/923 — Within the 31 days (Day 0-30) after the fourth dose phase
Teething (Gastrointestinal disorders) | 115/2769 | 46/923 — Within the 31 days (Day 0-30) after the fourth dose phase
Pain (General disorders) | 2419/3088 | 819/1016 — During the 4-day (Day 0-3) post primary vaccination course
Redness (General disorders) | 2052/3088 | 691/1016 — During the 4-day (Day 0-3) post primary vaccination course
Swelling (General disorders) | 1707/3088 | 568/1016 — During the 4-day (Day 0-3) post primary vaccination course
Drowsiness (General disorders) | 2418/3088 | 804/1015 — During the 4-day (Day 0-3) post primary vaccination course
Fever (General disorders) | 1434/3089 | 463/1015 — During the 4-day (Day 0-3) post primary vaccination course
Irritability (General disorders) | 2740/3088 | 926/1015 — During the 4-day (Day 0-3) post primary vaccination course
Loss of appetite (General disorders) | 1764/3088 | 609/1015 — During the 4-day (Day 0-3) post primary vaccination course
Pain (General disorders) | 1319/2528 | 494/832 — During the 4-day (Day 0-3) post-vaccination period following the fourth dose
Redness (General disorders) | 1213/2528 | 463/833 — During the 4-day (Day 0-3) post-vaccination period following the fourth dose
Swelling (General disorders) | 936/2526 | 334/832 — During the 4-day (Day 0-3) post-vaccination period following the fourth dose
Increase in limb circumference (General disorders) | 1489/2769 | 503/923 — During the 4-day (Day 0-3) post-vaccination period following the fourth dose
Drowsiness (General disorders) | 1088/2526 | 381/830 — During the 4-day (Day 0-3) post-vaccination period following the fourth dose
Fever (General disorders) | 341/2527 | 134/831 — During the 4-day (Day 0-3) post-vaccination period following the fourth dose
Irritability (General disorders) | 1482/2526 | 534/830 — During the 4-day (Day 0-3) post-vaccination period following the fourth dose
Loss of appetite (General disorders) | 825/2526 | 287/830 — During the 4-day (Day 0-3) post-vaccination period following the fourth dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.